CLINICAL TRIAL: NCT00931528
Title: A Randomized, Double-blind, Placebo-controlled Phase III Trial to Evaluate the Effectiveness of a Phosphodiesterase 5 Inhibitor, Tadalafil, in Prevention of Erectile Dysfunction in Patients Treated With Radiotherapy for Prostate Cancer
Brief Title: Tadalafil in Preventing Erectile Dysfunction in Patients With Prostate Cancer Treated With Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RTOG 0831; CDR0000647146; NCI-2011-01934 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer; Sexual Dysfunction
Keywords: sexual dysfunction; stage IIB prostate cancer; stage IIA prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Experimental): Tadalafil
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tadalafil — Beginning ≤ 7 days after the start of radiotherapy, patients receive oral tadalafil 5mg once daily for 24 weeks.
  Arms: Tadalafil
Other: Placebo — Beginning ≤ 7 days after the start of radiotherapy, patients receive oral placebo once daily for 24 weeks.
  Arms: Placebo

SUMMARY:
RATIONALE: Tadalafil may help prevent erectile dysfunction (ED) in patients with prostate cancer that has been treated with radiation therapy. It is not yet known whether tadalafil is more effective than a placebo in preventing erectile dysfunction.

PURPOSE: This randomized phase III trial is studying tadalafil to see how well it works compared with a placebo in preventing erectile dysfunction in patients with prostate cancer treated with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether tadalafil maintains spontaneous (off-drug) erectile function, as measured by the International Index of Erectile Function (IIEF) as compared to placebo at weeks 28-30 after initiation of radiotherapy in patients with prostate cancer.

Secondary

* Determine the difference in spontaneous (off-drug) erectile function between tadalafil and placebo at 1 and 2 years.
* Determine the difference in overall sexual function as measured by the IIEF between tadalafil and placebo at weeks 28-30 and at 1 and 2 years.
* Determine differences in patient and partner overall sexual satisfaction as measured by the Sexual Adjustment Questionnaire (SAQ) between tadalafil and placebo at weeks 28-30 and at 1 and 2 years.
* Determine differences in patient and partner marital adjustment as measured by Locke's Marital Adjustment Test (LMAT) between tadalafil and placebo at weeks 28-30 and at 1 and 2 years.
* Determine associations between patient and partner overall sexual satisfaction as measured by SAQ and patient and partner marital adjustment as measured by LMAT at weeks 28-30 and at 1 and 2 years.
* Determine patient-related factors (i.e., age, pretreatment sexual response, tobacco use, and comorbidities) that may predict response to tadalafil therapy at weeks 28-30 and at 1 and 2 years.
* Determine the difference in adverse events between tadalafil and placebo as assessed by Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 criteria.

Tertiary

* Characterization of preference and erectile function among patients who choose to stay on (or if on placebo, to start) tadalafil, a phosphodiesterase type 5 (PDE5) inhibitor other than tadalafil, a non-PDE5-inhibitor erectile aide, or no PDE5 inhibitor or erectile aide at 28-30 weeks and at 1 and 2 years.
* Identification of radiotherapy factors (i.e., modality, prescribed total dose, planning target volume margin, penile bulb dose-volume parameters) associated with erectile function.
* Evaluation of the number of patients screened for eligibility, the number eligible that are presented the study, the number who refuse, and the number who are accrued.

OUTLINE: This is a multicenter study. Patients are stratified according to age (≤ 65 years vs > 65 years) and radiotherapy treatment (external beam radiation therapy vs brachytherapy*). Patients are randomized to 1 of 2 treatment arms.

Note: * Radiotherapy start date for brachytherapy patients is the date of the procedure.

All patients undergo either external beam radiotherapy alone to the prostate ± seminal vesicles only or low-dose rate permanent brachytherapy alone.

* Arm I: Beginning ≤ 7 days after the start of radiotherapy, patients receive oral tadalafil once daily for 24 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Beginning ≤ 7 days after the start of radiotherapy, patients receive oral placebo once daily for 24 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete the International Index of Erectile Function (IIEF), the Sexual Adjustment Questionnaire (SAQ), the Locke's Marital Adjustment Test (LMAT) (if applicable), and the Expanded Prostate Cancer Index Composite Sexual Medications and Devices Evaluations Supplement questionnaires periodically. Partners or spouses complete the SAQ-Partner, LMAT (if applicable), and IIEF questionnaires periodically.

After completion of study treatment, patients are followed at 28-30 weeks, and annually for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stage T1b-T2b (AJCC, 6th ed.) adenocarcinoma of the prostate within 6 months of registration
2. Clinically negative lymph nodes as established by imaging (pelvic ± abdominal CT or MR), nodal sampling, or dissection within 3 months prior to registration. Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are ≤ 1.5 cm. Lymph node assessment is optional, and at investigator discretion, for patients with Gleason Score <7.
3. No evidence of bone metastases (M0) on bone scan within 3 months prior to registration. Equivocal bone scan findings are allowed if plain films are negative for metastasis. Bone metastases assessment is optional, and at investigator discretion, for patients with Gleason Score <7.
4. Baseline serum prostatic specific antigen (PSA) value performed with an FDA-approved assay (e.g., Abbott, Hybritech) within 3 months prior to registration.

   -4.1 Any of the following combinations of factors (NOTE: tumor found in 1 or both lobes on biopsy, but not palpable, will not alter T stage):
   * T1b-T2b disease, Gleason Score <7 and serum total PSA that is <20 ng/ml or
   * T1b-T2b disease, Gleason Score ≥7 and PSA that is <15 ng/ml
5. Serum total testosterone level prior to the initiation of radiation therapy (RT) within normal range according to institutional guidelines
6. Zubrod Performance Status 0 or 1 (Appendix III)
7. Age ≥ 18 years
8. Treatment that will consist of either external beam RT alone to the prostate ± seminal vesicles only at a dose between 75 Gy and 79.2 Gy or brachytherapy alone (NOTE: treatment with combined external RT and brachytherapy excludes patient participation)
9. Pretreatment (before starting prostate cancer treatment) erectile function as measured by IIEF Question 1, "How often were you able to get an erection during sexual activity?" - with responses of:

   * "sometimes (about half the time)" [response 3] or
   * "most times (much more than half the time)" [response 4] or
   * "almost always/always" [response 5]
10. History of prior tadalafil use: Document usual dosage per sexual encounter, date of last dose, and patient's response (No; Yes-Unsatisfactory Response; Yes-Satisfactory Response). Regardless of past experience, the patient is eligible if he agrees to adhere to protocol and take only tadalafil or placebo prescribed on study.
11. Although patients with partners are targeted for recruitment, patients without partners or without partners willing to participate are eligible. Patients (and spouses/partners, if willing to participate) must be able to provide study-specific informed consent.

Exclusion Criteria:

1. The patient's participation in another medical research study that involves the treatment of ED
2. Previous or concomitant invasive cancer (American Joint Committee on Cancer [AJCC] Stage >0), other than localized basal cell or squamous cell skin carcinoma (AJCC Stage 0-II), or a hematological malignancy (e.g., leukemia, lymphoma, myeloma) unless continually disease free for at least 5 years
3. History of myocardial infarction within the last year
4. Heart failure in the last 6 months
5. Uncontrolled arrhythmias, hypotension (<90/50mm Hg), or uncontrolled hypertension (>170/100 mm Hg)
6. Stroke within the last 6 months
7. Use of luteinizing hormone-releasing hormone (LHRH) agonist androgen suppression (e.g., Lupron, Zoladex), anti-androgen (e.g., Casodex, Eulexin, Nilandron), or estrogenic (e.g., diethylstilbestrol) agents within the last 6 months
8. Current use of any organic nitrate or as needed nitrates (e.g., use of nitroglycerin)
9. Current use of cimetidine, ketoconazole, itraconazole, erythromycin, or ritonavir
10. Known moderate to severe renal insufficiency or end-stage renal disease
11. Known severe hepatic impairment
12. Use of mechanical (vacuum) devices, intracorporeal, intraurethral, topical, or oral (sildenafil, tadalafil, vardenafil) agents as therapy for ED or supplements to enhance sexual function within 5-7 days prior to the start of RT. Patients who discontinue these therapies remain eligible if they can meet eligibility criteria
13. Pretreatment (before starting prostate cancer treatment) ED as measured by IIEF Question 1, "How often were you able to get an erection during sexual activity?" - with responses of:

    * "no sexual activity" [response 0] or
    * "almost never/never" [response 1] or
    * "a few times (much less than half the time)" [response 2]
14. Prior penile implant or history of bilateral orchiectomy
15. Prior prostatectomy, prostatic cryosurgery or high-intensity focused ultrasound (HIFU), radionuclide prostate brachytherapy, or chemotherapy for prostate cancer
16. Prior or anticipated combined external RT and brachytherapy
17. Prior or anticipated external RT to the pelvic ± para-aortic lymph nodes
18. Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immunocompromised patients.
19. Anatomical genital abnormalities or concurrent conditions that in the estimation of the physician would prohibit sexual intercourse or prevent study completion
20. Major medical or psychiatric illness which, in the opinion of the investigator, would prevent completion of treatment or would interfere with follow-up

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Watkins Bruner, RN, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (192):
- United States (183):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Enloe Medical Center, Chico, California
  - Saint Agnes Medical Center, Fresno, California
  - Veterans Administration Long Beach Medical Center, Long Beach, California
  - Northridge Hospital Medical Center, Northridge, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Radiological Associates of Sacramento, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - UCSF-Mount Zion, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center, Vallejo, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Broward Health North, Deerfield Beach, Florida
  - University of Florida, Gainesville, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Cancer Specialists of North Florida-Southside, Jacksonville, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida-Baptist South, Jacksonville, Florida
  - Cancer Specialists of North Florida-Beaches, Jacksonville Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Cancer Specialists of North Florida-Saint Augustine, Saint Augustine, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - IU Health Bloomington, Bloomington, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - IU Health Goshen Center for Cancer Care, Goshen, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Clinic CCOP, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - Tate Cancer Center, Glen Burnie, Maryland
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - McLaren-Flint, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Good Samaritan Hospital, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Concord Hospital, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - Southside Hospital, Bay Shore, New York
  - Lourdes Hospital, Binghamton, New York
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - The Coleman Radiation Center-Carteret General Hospital, Morehead City, North Carolina
  - CarolinaEast Health System-Medical Center, New Bern, North Carolina
  - South Atlantic Radiation Oncology, Supply, North Carolina
  - Coastal Carolina Radiation Oncology, Wilmington, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Flower Hospital, Sylvania, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Academic Urology Prostate Center, King of Prussia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology-Denton South, Denton, Texas
  - The Klabzuba Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - West Texas Cancer Center, Odessa, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Virginia, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Mason CCOP, Seattle, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Appleton Medical Center, Appleton, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - CHUQ - Pavilion Hotel-Dieu de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Derived] Pisansky TM, Pugh SL, Greenberg RE, Pervez N, Reed DR, Rosenthal SA, Mowat RB, Raben A, Buyyounouski MK, Kachnic LA, Bruner DW. Tadalafil for prevention of erectile dysfunction after radiotherapy for prostate cancer: the Radiation Therapy Oncology Group [0831] randomized clinical trial. JAMA. 2014 Apr 2;311(13):1300-7. doi: 10.1001/jama.2014.2626. PMID 24691606

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 121 | 121
Completed | 80 (Subjects with data available for the primary analysis are considered to have completed the study.) | 61 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 41 | 60
Not completed — Protocol Violation | 9 | 12
Not completed — Withdrawal by Subject | 4 | 12
Not completed — Lost to Follow-up | 6 | 13
Not completed — Assessment outside of Time Frame | 22 | 23

BASELINE CHARACTERISTICS:
Population: All randomized eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 112 | 109 | 221
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 80] | 63 [48 to 79] | 63 [45 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 112 | 109 | 221

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Maintaining Spontaneous (Off-drug) Erectile Function (EF) at Weeks 28-30 After Initiation of Radiation Therapy (RT)
Description: EF is measured by Question 1 of the International Index of Erectile Function (IIEF). The IIEF is a validated 15-item for measuring patient-reported erectile function. Question 1 asks "How often were you able to get an erection during sexual activity?" Responses ranged from 0=no sexual activity, to 5=Almost always or always. Higher scores indicated better functioning. All patients have erectile function prior to initiation of RT, indicated by a score of 3, 4, or 5 on IIEF Q1. Patients with a lower IIEF Q1 score at weeks 28-30 than at baseline will have less erectile function and be categorized as nonresponders. Patients with similar or improved erectile function will be categorized as responders (maintaining). Patient-related predictors of at erectile function at this time point are also reported with this outcome measure.
Time Frame: Baseline and 30 weeks from the start of radiation therapy
Population: All randomized eligible patients with IIEF at both baseline and 30 week time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tadalafil: Beginning ≤ 7 days after the start of radiotherapy, patients receive oral tadalafil once daily for 24 weeks.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 80 | 61
percentage of participants | 79 [70 to 88] | 74 [63 to 85]
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Sample size calculations were based on the hypothesis that the use of tadalafil would statistically significant increase the proportion of patients maintaining spontaneous erectile function compared to the use of placebo. Based on a 2-sided Fisher exact test with alpha=0.05, 91 patients/arm would provide 80% statistical power to detect an increase from 20% to 40% in spontaneous erectile response at weeks 28-30. Although designed for the Fisher exact test, Chi-square was used and reported; Test type: Superiority or Other; p = 0.49, Chi-squared; Difference in percentages = 5, 95% CI 2-sided [1 to 9]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX vs. N0)] were retained in the model. (Dropped: ethnicity, Zubrod, T stage, prostate-specific antigen (PSA).) The results for each explanatory variable are reported separately. Treatment arm is reported here; Test type: Superiority; p = 0.2386, Regression, Logistic
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX vs. N0)] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, T stage, PSA.)The results for each explanatory variable are reported separately. RT method is reported here; Test type: Superiority; p = 0.7908, Regression, Linear
Statistical Analysis 4: Comparison: Tadalafil vs Placebo; Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX vs. N0)] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, T stage, PSA.) The results for each explanatory variable are reported separately. Age is reported here; Test type: Superiority; p = 0.0467, Regression, Logistic
Statistical Analysis 5: Comparison: Tadalafil vs Placebo; Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX vs. N0)] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, T stage, PSA.) The results for each explanatory variable are reported separately. N Stage is reported here; Test type: Superiority; p = 0.0068, Regression, Logistic

2. Secondary Outcome: Percentage of Patients Maintaining Spontaneous (Off-drug) EF at Years 1 and 2 After Initiation of RT
Description: The International Index of Erectile Function (IIEF) is a validated 15-item for measuring patient-reported erectile function. Question 1 asks "How often were you able to get an erection during sexual activity?" Responses ranged from 0=no sexual activity, to 5=Almost always or always. Higher scores indicated better functioning. All patients have erectile function prior to initiation of RT, indicated by a score of 3, 4, or 5. Patients with a lower IIEF Q1 score at weeks 28-30 than at baseline will have less erectile function and be categorized as nonresponders. Patients with similar or improved erectile function will be categorized as responders (maintaining). Patient-related predictors of at erectile function at Years 1 and 2 are also reported with this outcome measure.
Time Frame: Baseline, 1 and 2 years from the start of tadalafil or placebo
Population: All randomized eligible patients with IIEF at both baseline and corresponding time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 109 | 108
percentage of participants
  Year 1: number analyzed (Participants) | 54 | 49
  Year 1 | 72.2 [60.3 to 84.1] | 71.4 [58.7 to 84.1]
  Year 2: number analyzed (Participants) | 57 | 49
  Year 2 | 68.4 [56.3 to 80.5] | 63.3 [49.8 to 76.8]
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Year 1; Test type: Superiority; p = 0.93, Chi-squared; 2-sided significance level = 0.05
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; Year 2; Test type: Superiority; p = 0.58, Chi-squared; 2-sided significance level = 0.05
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; Year 1: Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [none] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, N stage, T stage, PSA.) The results for each explanatory variable are reported separately. Treatment arm is reported here; Test type: Superiority; p = 0.9501, Regression, Logistic
Statistical Analysis 4: Comparison: Tadalafil vs Placebo; Year 1: Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [none] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, N stage, T stage, PSA.) The results for each explanatory variable are reported separately. RT method is reported here; Test type: Superiority; p = 0.1020, Regression, Logistic
Statistical Analysis 5: Comparison: Tadalafil vs Placebo; Year 1: Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [none] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, N stage, T stage, PSA.) The results for each explanatory variable are reported separately. Age is reported here; Test type: Superiority; p = 0.1855, Regression, Logistic
Statistical Analysis 6: Comparison: Tadalafil vs Placebo; Year 2: Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX)] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, T stage, PSA.) The results for each explanatory variable are reported separately. Treatment arm is reported here; Test type: Superiority; p = 0.5739, Regression, Logistic
Statistical Analysis 7: Comparison: Tadalafil vs Placebo; Year 2: Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX)] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, T stage, PSA.) The results for each explanatory variable are reported separately. RT method is reported here; Test type: Superiority; p = 0.0422, Regression, Logistic
Statistical Analysis 8: Comparison: Tadalafil vs Placebo; Year 2: Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX)] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, T stage, PSA.) The results for each explanatory variable are reported separately. Age is reported here; Test type: Superiority; p = 0.5237, Regression, Logistic
Statistical Analysis 9: Comparison: Tadalafil vs Placebo; Year 2: Logistic regression using generalized estimating equations was performed modeling the probability of non-responders. Only treatment arm (Placebo vs. Tadalafil), age (> 65 vs. other), RT method (External RT vs. brachytherapy), and significant pretreatment characteristics [N stage (NX)] were retained in the model. (Dropped pretreatment characteristics: ethnicity, Zubrod, T stage, PSA.) The results for each explanatory variable are reported separately. N Stage is reported here; Test type: Superiority; p = 0.4770, Regression, Logistic

3. Secondary Outcome: Overall Sexual Function as Measured by Change From Baseline in the International Index of Erectile Function (IIEF)
Description: The IIEF is a validated 15-item for measuring patient-reported erectile function. A score of 0-5 is given to each of the 15 questions that examine 5 main domains of male sexual function: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Domain scores are the sum of each item. The erectile function domain has 5 items with a score range of 1-30, orgasmic function has 2 items with a score range of 0-10, sexual desire has 2 items with a score range of 0-10, intercourse satisfaction has 3 items with a score range of 0-15, and overall satisfaction has 2 items with a score range of 2-10. Total score ranges from 0-70, with higher scores indicated better functioning. Change from baseline is calculated by subtracting baseline score from score at the time point of interest.
Time Frame: Baseline, week 30, and years 1 and 2 from start of treatment
Population: Eligible patients with IIEF at baseline and corresponding time points.
Measure: Mean (Standard Deviation); unit: change in total IIEF
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 109 | 108
change in total IIEF
  Week 30: number analyzed (Participants) | 70 | 58
  Week 30 | -8.2 (15.4) | -9.0 (17.0)
  Year 1: number analyzed (Participants) | 46 | 45
  Year 1 | -9.5 (14.8) | -10.5 (18.4)
  Year 2: number analyzed (Participants) | 49 | 45
  Year 2 | -9.7 (15.7) | -14.1 (20.1)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Week 30; Test type: Superiority; p = 0.97, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; Year 1; Test type: Superiority; p = 0.99, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; Year 2; Test type: Superiority; p = 0.24, t-test, 2 sided; Significance level = 0.05

4. Secondary Outcome: Overall Patient Sexual Satisfaction as Measured by Change From Baseline in the Sexual Adjustment Questionnaire (SAQ) Score
Description: The Sexual Adjustment Questionnaire (SAQ) is a 20-item questionnaire with an overall score range between 8 and 100 including the following domains: desire, ranging between 5 and 30; dysfunction, 0 and 25; activity, 0 and 10; satisfaction, 1 and 10; and fatigue, 1 and 5. The change in SAQ score is calculated by subtracting the baseline score from the follow-up score. A positive change indicates an improvement in sexual well-being.
Time Frame: Baseline, week 30 and years 1 and 2 after the start of treatment
Population: Eligible patients with data at baseline and corresponding time point
Measure: Mean (Standard Deviation); unit: change in SAQ score
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 63 | 51
change in SAQ score
  Week 30: number analyzed (Participants) | 47 | 35
  Week 30 | -2.0 (11.3) | -2.9 (8.0)
  Year 1: number analyzed (Participants) | 36 | 24
  Year 1 | -3.7 (9.7) | -4.9 (9.9)
  Year 2: number analyzed (Participants) | 31 | 28
  Year 2 | -3.4 (9.3) | -4.6 (14.8)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Week 30; Test type: Superiority; p = 0.70, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; Year 1; Test type: Superiority; p = 0.65, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; Test type: Superiority; p = 0.72, t-test, 2 sided; Significance level = 0.05

5. Secondary Outcome: Overall Partner Sexual Satisfaction as Measured by Change From Baseline in the Sexual Adjustment Questionnaire-Partner (SAQ-P) Score
Description: The SAQ-P is an 18-item questionnaire with an overall score range between 0 and 90 including the following domains: desire, dysfunction, activity, satisfaction, and fatigue. The change in SAQ score is calculated by subtracting the baseline score from the follow-up score. A positive change indicates an improvement in sexual well-being.
Time Frame: Baseline, week 30 and years 1 and 2 after the start of treatment
Population: Consenting partners of randomized eligible patients with data at baseline and corresponding time point
Measure: Mean (Standard Deviation); unit: change in SAQ score
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 42 | 40
change in SAQ score
  Week 30: number analyzed (Participants) | 27 | 20
  Week 30 | -4.9 (7.5) | -1.8 (8.2)
  Year 1: number analyzed (Participants) | 21 | 20
  Year 1 | -3.9 (6.4) | -2.5 (7.1)
  Year 2: number analyzed (Participants) | 18 | 16
  Year 2 | 1.5 (5.5) | 5.1 (9.6)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Week 30; Test type: Superiority; p = 0.14, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; Year 1; Test type: Superiority; p = 0.64, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; Year 2; Test type: Superiority; p = 0.18, t-test, 2 sided; Significance level = 0.05

6. Secondary Outcome: Patient Marital Adjustment as Measured by the Locke's Marital Adjustment Test
Description: The Locke Marital Adjustment Test (LMAT) is a 16-item questionnaire with scores ranging from 48 to 138 for participants. Higher scores indicate greater sexual function, sexual wellbeing, or marital adjustment. The change in LMAT score is calculated by subtracting the baseline score from the follow-up score.
Time Frame: Baseline, week 30 and years 1 and 2 after the start of treatment
Population: Eligible patients with data at baseline and time point of interest.
Measure: Mean (Standard Deviation); unit: change in LMAT score
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 61 | 60
change in LMAT score
  Week 30: number analyzed (Participants) | 35 | 29
  Week 30 | -3.5 (7.7) | -2.6 (10.4)
  Year 1: number analyzed (Participants) | 22 | 23
  Year 1 | -1.9 (7.2) | -1.9 (6.3)
  Year 2: number analyzed (Participants) | 27 | 27
  Year 2 | -1.3 (9.87) | -1.4 (5.4)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Week 30; Test type: Superiority; p = 0.67, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; Year 1; Test type: Superiority; p = 0.98, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; Year 2; Test type: Superiority; p = 0.96, t-test, 2 sided; Significance level = 0.05

7. Secondary Outcome: Partner Marital Adjustment as Measured by the Locke's Marital Adjustment Test
Description: as for outcome 6
Time Frame: Baseline, week 30 and years 1 and 2 after the start of treatment
Population: Consenting spouses of randomized, eligible patients with data at baseline and time point of interest
Measure: Mean (Standard Error); unit: change in LMAT score
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 34 | 27
change in LMAT score
  Week 30: number analyzed (Participants) | 19 | 12
  Week 30 | -1.5 (6.3) | -2.6 (6.4)
  Year 1: number analyzed (Participants) | 16 | 12
  Year 1 | -2.3 (5.1) | 1.2 (7.3)
  Year 2: number analyzed (Participants) | 13 | 9
  Year 2 | -2.8 (5.8) | -4.7 (7.1)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Week 30; Test type: Superiority; p = 0.86, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; Year 1; Test type: Superiority; p = 0.93, t-test, 2 sided; Significance level = 0.05
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; Year 2; Test type: Superiority; p = 0.52, t-test, 2 sided; Significance level = 0.05

8. Other Pre Specified Outcome: Radiotherapy Factors Associated With Spontaneous (Off-drug) EF at Weeks 28-30 and Years 1 and 2 After Initiation of RT
Time Frame: Baseline, week 30 and years 1 and 2 after the start of treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Patient Follow-up Treatment for Erectile Dysfunction at Weeks 28-30 and Years 1 and 2 After Initiation of RT
Time Frame: Baseline, week 30 and years 1 and 2 after the start of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse event (AE) data is reported for eligible patients with adverse event data. Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events.
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 3/111 | 4/108
Other Adverse Events (participants affected / at risk) | 85/111 | 76/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tadalafil (N=111) | Placebo (N=108)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Investigations - Other (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Visceral arterial ischemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tadalafil (N=111) | Placebo (N=108)
Diarrhea (Gastrointestinal disorders) | 18 | 10
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 7 | 2
Fatigue (General disorders) | 30 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Headache (Nervous system disorders) | 9 | 4
Cystitis noninfective (Renal and urinary disorders) | 7 | 10
Renal and urinary disorders - Other (Renal and urinary disorders) | 22 | 21
Urinary frequency (Renal and urinary disorders) | 55 | 50
Urinary retention (Renal and urinary disorders) | 17 | 19
Urinary tract pain (Renal and urinary disorders) | 15 | 14
Urinary urgency (Renal and urinary disorders) | 36 | 22
Ejaculation disorder (Reproductive system and breast disorders) | 7 | 6
Erectile dysfunction (Reproductive system and breast disorders) | 34 | 31
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 6 | 0
Hypertension (Vascular disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
The protocol endpoint "Patient-related predictors of erectile function" refers to modeling of the first two outcome measures, and is therefore reported as additional statistical analyses for those outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.